CLINICAL TRIAL: NCT03934021
Title: Gut Microbiota in Acute Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. IP Yiu Ming Bonaventure, Clinical Tutor, Chinese University of Hong Kong
Other Study IDs: crec 2016.545
Record Dates: First submitted 2019-04-25; First posted 2019-05-01 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Stroke, Acute; Stroke, Ischemic; Microbiome; Atherosclerosis Cerebral
Keywords: Stroke; Ischemic stroke; microbiome; atherosclerotic
MeSH Terms: conditions — Stroke; Ischemic Stroke; Intracranial Arteriosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stools samples will be stored at -80 degrees Celsius within 24 hours after collection. 16S rRNA gene amplicons will be obtained through DNA extraction, PCR amplification and purification using available kits. After pyrosequencing, sequences will be analysed using mother pipeline and grouped into operational taxonomic units and classified using GreenGenes. OTU based microbial diversity was estimated by calculating the nonparametric Shannon diversity index. Alpha diversity and abundance profiles will be used for downstream statistical and modeling analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute stroke patient group: Consecutive patients diagnosed with acute ischaemic stroke during hospitalization in Prince of Wales Hospital will be recruited.
  After an informed consent, stool will be collected from enrolled patients in their first bowel opening after hospitalization and stored in a freezer (-80 degree Celsius) within 24 hours for analysis. If a subject develops constipation, stool sampling will be facilitated by stool softener or laxatives. Stools samples will be stored at -80 degrees Celsius within 24 hours once it is collected.
  Subjects will be followed up at 3 and 6 months after trial entry. NIHSS and mRS will be performed at each visit. Stool sample collection will be repeated in 6 months visit only.
- Control group: Age and disease matched subjects will be invited to join the study as the control. Stool will also be collected for the comparison of gut microbiota with acute stroke patients to look for evidence of gut dysbiosis in acute stroke. We shall match the control cohort with the stroke cohort in terms of age, gender, smoking status, medical co-morbidities including hypertension, hyperlipidaemia, diabetes, (atrial fibrillation), use of medications in particular metformin, proton pump inhibitors and aspirin.

SUMMARY:
This study is to find out the significance of gut-microbiota in acute stroke patients, including their neurological, radiological outcomes as well as their stroke mechanisms.

DETAILED DESCRIPTION:
Patients who suffered from acute stroke and in hospitalization in Prince of Wales Hospital will be recruited in the study.

After the informed consent, their first bowel opening will be collected for storage. They will also receive assessment by the stroke team at 3 and 6 months to determine their outcomes (NIHSS and mRS). Clinically and radiologically parameters including their degree of disability, imaging findings will also be collected to determine whether there are any correlations with the stool microbiota composition against matched individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as acute ischaemic stroke
2. Aged 18 or above Chinese
3. Radiological evidence of acute ischaemic stroke by Computed tomography (CT) or magnetic resonance imaging (MRI) brain.

Exclusion Criteria:

1. Patient with symptoms and signs suggestive of alternative diagnoses,
2. Evidence of intracerebral haemorrhage,
3. Absence of DWI evidence of acute ischaemic infarct,
4. Pregnancy,
5. Evidence of gastrointestinal infection/ inflammation/ obstruction
6. History of partial or total resection of small or large bowel, as well as gut re-anastomosis,
7. Use of antibiotics within 2 weeks prior to symptoms onset,
8. Gastrointestinal malignancy
9. Any hospitalization within 3 months before recruitment
10. Institutionalized patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients diagnosed with acute ischaemic stroke during hospitalization in PWH will be recruited. Eligibility will be determined through a checklist of inclusion and exclusion criteria. Control group will be recruited from medical out patient clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The composition of gut-microbiota contributing neurological outcome between groups | 31 Dec, 2020
  Gene sequencing of the 16S rRNA on the stool samples are performed to identify the microbes down to genus level, as well as the microbrobiota diversity and relative abundance. And stroke etiology classified by TOAST Classification and disability indices (NIHSS & mRS at baseline, 3 month & 6 month) will be recorded.

SECONDARY OUTCOMES:
The composition of gut-mircobiota contributing radiological finding between groups | 31 Dec, 2020
  Gene sequencing of the 16S rRNA on the stool samples are performed to identify the microbes down to genus level, as well as the microbrobiota diversity and relative abundance. All patients who received a plain CT brain & MRI for the diagnosis of stroke will be reviewed. Infarct volume in DWI, MR angiography abnormalities, presence of microbleed and/or haemorrhagic transformation will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Yiu Ming Bonaventure IP, MRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided